CLINICAL TRIAL: NCT02562521
Title: A Smoking Cessation Intervention for Yale Dining Employees
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1411014980
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoking Cessation Treatment (Experimental): The intervention will consist of Contingency management (CM) in conjunction with effective first line pharmacotherapy (dual nicotine replacement therapy [NRT] or varenicline) and brief counseling to rapidly induce cessation and to maintain abstinence long term. Pharmacotherapy will be flexible. Participants will also be given the option of receiving additional behavioral support by being referred to the CT Quitline and using text or mobile phone apps for quitting.
  Interventions: Behavioral: Contingency management; Drug: Nicotine replacement therapy; Drug: Varenicline; Behavioral: Additional behavioral support
- Delayed Treatment Control (No Intervention): Participants in this arm will be offered the Smoking Cessation Treatment 6 weeks later

INTERVENTIONS:
Behavioral: Contingency management — Participants in the intervention group will receive a tailored intervention that utilizes contingency management in which they receive monetary rewards for reducing or quitting smoking.
  Arms: Smoking Cessation Treatment
Drug: Nicotine replacement therapy — Participants have the option of using nicotine patch in combination with nicotine gum or lozenge
  Arms: Smoking Cessation Treatment
Drug: Varenicline — Individuals who do not respond initially to Nicotine Replacement Therapy will be offered varenicline as an alternative
  Arms: Smoking Cessation Treatment
Behavioral: Additional behavioral support — Based on interest, participants can be referred to a telephone quitline or receive access to mobile text messaging programs or app based smoking cessation support
  Other Names: telephone quit lines and mobile applications
  Arms: Smoking Cessation Treatment

SUMMARY:
The purpose of this study is to evaluate a smoking cessation program for employees at the Yale University dining hall. Two pilot dining halls and six paired dining halls (3 test and 3 control sites) will be offered a contingency management/pharmacotherapy smoking cessation intervention at the work site.

DETAILED DESCRIPTION:
The primary aim of this study is to test the effect of a smoking cessation intervention provided to Yale University dining hall employees on smoking quit rates and quit attempts at the end of six weeks of treatment. It is hypothesized that participants from the test site will have higher rates of smoking cessation and quit attempts compared to participants from the control site. In addition, this study will examine the number of participants who enroll in the smoking cessation program who successfully quit smoking at 6 months.

There will be 3 test sites and 3 control sites in this study (broken down into 3 pairs of test/control). Each test site will be matched to on a control site. Self-reported smoking status will be obtained for all participants in the test and control sites at 3 time points (baseline, 6 weeks and 6 months). The study start time for each pair will be delayed by 4-8 weeks for feasibility issues.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker
* Interested in receiving treatment for quitting smoking.
* Employed for more than 20 hours per week by one of the 7 residential college dining halls selected for inclusion in this study.
* English speaker.

Exclusion Criteria:

* None specified, other than failure to meet all inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie O'Malley, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Site Participants; Control Site Participants: Dining hall employees who were current smokers were invited to participate in a treatment research study. Participants in the test and control sites received the same treatment components with a time delay where the control site started treatment 6 weeks after the test site.
Period: Overall Study
Arm/Group | Test Site Participants | Control Site Participants
Started | 18 | 7
Completed | 18 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Dining hall employees who were current smokers were invited to participate in a treatment research study. Participants in the test and control sites received the same treatment components with a time delay where the control site started treatment 6 weeks after the test site.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Site Participants | Control Site Participants | Total
Number analyzed (Participants) | 18 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (13.3) | 43.2 (11.6) | 44.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 8 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 7 | 21
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 4 | 16
  White | 2 | 2 | 4
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Smoking Quit Attempt in the Prior Six Weeks
Description: A survey of dining hall employees will be used to determine the proportion of the dining hall employees who made a quit attempt in the prior six weeks in the treatment and delayed treatment control groups. Values present the proportion of dining hall employees who smoke who reported making a quit attempt.
Time Frame: 6 weeks
Population: These analyses are conducted for the subset of dining hall employees who reported being smokers.
Measure: Count of Participants; unit: Participants
Groups:
- Smoking Cessation Treatment: The intervention will consist of Contingency management (CM) in conjunction with effective first line pharmacotherapy (dual nicotine replacement therapy [NRT] or varenicline) and brief counseling to rapidly induce cessation and to maintain abstinence long term. Pharmacotherapy will be flexible. Participants will also be given the option of receiving additional behavioral support by being referred to the CT Quitline and using text or mobile phone apps for quitting.
  Contingency management: Participants in the intervention group will receive a tailored intervention that utilizes contingency management in which they receive monetary rewards for reducing or quitting smoking.
  Nicotine replacement therapy: Participants have the option of using nicotine patch in combination with nicotine gum or lozenge
  Varenicline: Individuals who do not respond initially to Nicotine Replacement Therapy will be offered varenicline as an alternative
  Additional behavioral support: Based on interest,
Arm/Group | Smoking Cessation Treatment | Delayed Treatment Control
Number analyzed (Participants) | 15 | 8
Participants | 10 | 1

2. Primary Outcome: Number of Participants Who Quit Smoking for at Least 24 Hours in the Prior Six Weeks
Description: A survey of dining hall employees will be used to determine the proportion of the dining hall employees who quit smoking for at least 24 hours in the prior six weeks in the treatment and delayed treatment control groups. Values present the number of individuals who report quitting successfully for at least 24 hours among individuals who reported smoking.
Time Frame: 6 weeks
Population: These analyses are conducted for the subset of dining hall employees who reported being smokers.
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Treatment | Delayed Treatment Control
Number analyzed (Participants) | 15 | 8
Participants | 8 | 1

3. Secondary Outcome: Number of Participants Who Quit Smoking at 2 Months
Description: Smoking cessation is operationally defined as successfully quitting smoking at 2 months measured with TLFB (a standardized, validated, and reliable experimenter-administered rating scale that will be used to obtain quantity and frequency estimates of smoking) and confirmed with expired breath carbon monoxide reading (CO less than or equal to 4 parts per million).
Time Frame: Month 2
Population: These analyses are conducted for the subset of dining hall employees who enrolled in the treatment program. Results are combined across the treatment and delayed control groups during the follow-up period because both groups received the same treatment components so we did not differentiate outcomes between arm/group during the follow-up period.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants Enrolled in Treatment: All participants who enrolled in treatment in either the intervention condition or delayed treatment control were followed after treatment to determine smoking cessation outcomes.
Arm/Group | All Participants Enrolled in Treatment
Number analyzed (Participants) | 25
Participants | 2

4. Secondary Outcome: Number of Participants Who Quit Smoking at 3 Months
Description: Smoking cessation is operationally defined as successfully quitting smoking at 3 months measured with TLFB (a standardized, validated, and reliable experimenter-administered rating scale that will be used to obtain quantity and frequency estimates of smoking) and confirmed with expired breath carbon monoxide reading (CO less than or equal to 4 parts per million).
Time Frame: Month 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants Enrolled in Treatment
Number analyzed (Participants) | 25
Participants | 1

5. Secondary Outcome: Number of People Who Quit Smoking at 4 Months
Description: Smoking cessation is operationally defined as successfully quitting smoking at 4 months measured with TLFB (a standardized, validated, and reliable experimenter-administered rating scale that will be used to obtain quantity and frequency estimates of smoking) and confirmed with expired breath carbon monoxide reading (CO less than or equal to 4 parts per million).
Time Frame: Month 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants Enrolled in Treatment
Number analyzed (Participants) | 25
Participants | 4

6. Secondary Outcome: Number of People Who Quit Smoking at 5 Months
Description: Smoking cessation is operationally defined as successfully quitting smoking at 5 months measured with TLFB (a standardized, validated, and reliable experimenter-administered rating scale that will be used to obtain quantity and frequency estimates of smoking) and confirmed with expired breath carbon monoxide reading (CO less than or equal to 4 parts per million).
Time Frame: Month 5
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants Enrolled in Treatment
Number analyzed (Participants) | 25
Participants | 2

7. Secondary Outcome: Number of People Who Quit Smoking at 6 Months
Description: Smoking cessation is operationally defined as successfully quitting smoking at 6 months measured with TLFB (a standardized, validated, and reliable experimenter-administered rating scale that will be used to obtain quantity and frequency estimates of smoking) and confirmed with expired breath carbon monoxide reading (CO less than or equal to 4 parts per million).
Time Frame: Month 6
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants Enrolled in Treatment
Number analyzed (Participants) | 25
Participants | 1

8. Secondary Outcome: Wisconsin Predicting Patient's Relapse Questionnaire
Description: Items from the Wisconsin Predicting Patient's Relapse questionnaire (WI-PREPARE) will be administered. This is a brief scale comprised of 7 items that assesses proneness to smoking relapse. Items are summed to create a total score. Total range=1-13 with higher scores indicating greater likelihood of smoking relapse.
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants Enrolled in Treatment
Number analyzed (Participants) | 25
units on a scale | 5.64 (1.96)

9. Secondary Outcome: Wisconsin Predicting Patient's Relapse Questionnaire
Description: as for outcome 8
Time Frame: Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants Enrolled in Treatment
Number analyzed (Participants) | 25
units on a scale | 4.80 (1.74)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the treatment period through 6 month follow-up.
Description: These analyses are conducted for the subset of dining hall employees who enrolled in the treatment program. Results are combined across the treatment and delayed control groups because both groups received the same treatment components so we did not differentiate outcomes or adverse events between arm/group.
Groups:
- All Participants Who Enrolled in Treatment: All participants who enrolled in treatment in either the intervention condition or delayed treatment control were followed after treatment to determine smoking cessation and adverse event outcomes because all participants ultimately received the same treatment components.
Arm/Group | All Participants Who Enrolled in Treatment
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No